CLINICAL TRIAL: NCT05408975
Title: Treatment of Word Finding Difficulties and Verbal Retrieval Deficits in Civilians Who Sustain a Chronic Traumatic Brain Injury With High Definition Transcranial Direct Current Stimulation
Brief Title: Treating Civilian Traumatic Brain Injury With High Definition Transcranial Direct Current Stimulation (ciTBI-HDtDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-231; 1K99DC020185-01A1 (NIH); 5K99DC020185-02 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Word Finding Difficulty; Acquired Brain Injury; Cognitive Change
Keywords: transcranial direct current stimulation; electroencephalography; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic; Anomia; Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 treatment arms: (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule.
  Additionally, after completing the initial active or sham treatment and 2-month follow-up testing sessions, all participants will be invited back for newly assigned treatment conditions, 20 minutes over 10 sessions and will be and re-evaluated at 2-months follow-up testing sessions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, assessors, and technicians interacting with participants will be blind to assigned conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active to Sham Transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive active stimulation. After completion of active stimulation, subjects will be assigned to sham stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation
- Sham to Active transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive sham stimulation. After completion of sham stimulation, subjects will be assigned to active stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Active Transcranial direct current stimulation — Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
  Other Names: tDCS; 1 milliamp tDCS; High definition tDCS; High definition transcranial direct current stimulator, Neuroelectrics Starstim tES, SN E20200930-10
Device: Sham Transcranial direct current stimulation — Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.

SUMMARY:
The purpose of the study is to test whether low level electric stimulation, called transcranial Direct Current Stimulation (tDCS), on the part of the brain (i.e., pre-supplementary motor area) thought to aid in memory will improve verbal retrieval in civilian (non-military, non-veteran) participants with histories of traumatic brain injuries. The primary outcome measures are neuropsychological assessments of verbal retrieval, and the secondary measures are neuropsychological assessments of other cognitive abilities and electroencephalography (EEG) measures. Additionally, the study will examine the degree to which baseline assessments of cognition, concussion history, structural brain imaging, and EEG predict responses to treatment over time, both on assessments administered within the intervention period and at follow-up.

DETAILED DESCRIPTION:
Using two treatment arms, the study will examine improvement of verbal retrieval and other cognitive deficits associated with remote traumatic brain injury by comparing (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule. Additionally, after completing the initial active or sham treatment and 2-month follow-up testing sessions, participants will be invited back for newly assigned treatment conditions, 20 minutes over 10 sessions and will be re-evaluated at 2-months follow-up testing sessions.

Civilians with histories of traumatic brain injuries and observed cognitive deficits will be randomly assigned to one of the two treatment arms (and re-assigned for the second round of intervention, as described above). Primary outcome verbal retrieval measures, secondary neuropsychological and electroencephalography (EEG) measures, and prescreening assessments for study concussion history and contraindications for treatment will be collected prior to being assigned to a treatment arm (i.e., baseline). Magnetic resonance imaging of the brain will be obtained only at the baseline assessment.

Primary outcome verbal retrieval measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected after treatment session 10 and one time following treatment competition (i.e., 2-months). For participants who complete the second round of intervention, primary outcome verbal memory measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected again after treatment session 10 and one time following competition of the second treatment (i.e., 2-months).

This study was funded by NIH/NIDCD under grant number [1K99DC020185]. Federal funding concluded on 11/30/2024.

ELIGIBILITY:
Inclusion Criteria: Participants are to be between the ages of 18-85, are non-military personnel and not veterans, and have had a traumatic brain injury (more than a year ago prior to study participation) that has led to a complaint of word finding difficulty since the brain injury, confirmed to represent a verbal retrieval deficit based on neuropsychological testing criteria. Traumatic brain injury must be in the mild to moderate range based on evaluation, including the Ohio State TBI Identification Method (administered by our research group). You must be fluent in speaking and reading English.

Exclusion Criteria:

* an implanted/electronic device, such as a pacemaker, metallic cranial or intracranial implant (e.g., ventriculoperitoneal shunt), or a neurostimulator (e.g., vagus nerve stimulator, spinal stimulator, deep brain stimulator, etc.).
* skull defects
* a history of a psychological or neurological disorder, including, dementia of any type, epilepsy or other seizure disorders, post-traumatic stress disorder, brain tumor, present drug abuse, stroke, blood vessel abnormalities in the brain, Parkinson's disease, Huntington's disease, or multiple sclerosis.
* inability to give informed consent
* currently pregnant
* not a native English speaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, MD, Principal Investigator — The University of Texas at Dallas
Locations (2):
- United States (2):
  - The University of Texas at Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Will share data upon request.

REFERENCES:
- [Result] Adhikari. A., Devora, P., Vintila, T., Mathews, A., Nguyen, B., Motes, M., LoBue, C., Cullum, C.M., Hart, J., Chiang, H.-S., B - 36 Investigating High-Definition Transcranial Direct Current Stimulation for Remediating Word Finding Difficulty in Civilians with a History of Chronic Traumatic Brain Injury: a Pilot Study, Archives of Clinical Neuropsychology, Volume 39, Issue 7, October 2024, Page 1126

RESULTS

PARTICIPANT FLOW:
Groups:
- Active to Sham Transcranial Direct Current Stimulation: Subjects in this arm were first randomly assigned to receive active stimulation. After completion of active stimulation, subjects were assigned to sham stimulation.
- Sham to Active Transcranial Direct Current Stimulation: Subjects in this arm were first randomly assigned to receive sham stimulation. After completion of sham stimulation, subjects were assigned to active stimulation.
Period: Baseline
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Immediately Post Phase 1 Intervention
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: 8 Weeks Post Phase 1 Intervention
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Immediately Post Phase 2 Intervention
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Period: 8 Weeks Post Phase 2 Intervention
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 47.7 (24.6) | 50 (15.6) | 48.6 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 3 | 2 | 5
The Controlled Oral Word Association Test [Mean (Standard Deviation); unit: items] — Evaluation of the Control Word Association Test. Metric: Total Number of Correct Items Generated for three different letters. Total Range 0 (minimum) - 200 (maximum). Larger numbers indicate better performance.
  items | 30.67 (7.23) | 30.5 (0.71) | 30.6 (5.13)
Category Fluency [Mean (Standard Deviation); unit: Total items] — Evaluation of Category Fluency. Metric: Total Number of Correct Items Generated for Animal. Total Range 0 (minimum) - 100 (maximum). Larger numbers indicate better performance.
  Total items | 18 (1.73) | 17 (0) | 17.6 (1.34)
The Boston Naming Test [Mean (Standard Deviation); unit: Total items] — Evaluation of the Boston Naming Test - 30 items. Metric: Total Number of Correct Items Generated. Total Range 0 (minimum) - 30 (maximum). Larger numbers indicate better performance.
  Total items | 26.67 (2.52) | 28 (0) | 27.2 (1.93)
Semantic Object Retrieval Test [Mean (Standard Deviation); unit: Total items] — Evaluation o Semantic Object Retrieval Test. Metric: Total Number of Correct Retrievals. Total Range 0 (minimum) - 32 (maximum). Larger numbers indicate better performance.
  Total items | 30.33 (1.53) | 30.5 (2.12) | 30.4 (1.52)
The Delis Kaplan Color Word Interference Test, naming [Mean (Standard Deviation); unit: Time- Seconds] — Evaluation of the Delis Kaplan Color Word Interference Test. Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 150 (maximum). Longer time indicates worse performance.
  Time- Seconds | 35.66666667 (5.131601439) | 41 (7.071067812) | 37.8 (5.85)
The Delis Kaplan Color Word Interference Test, reading [Mean (Standard Deviation); unit: Time - seconds] — Evaluation of the Delis Kaplan Color Word Interference Test. Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 150 (maximum). Longer time indicates worse performance.
  Time - seconds | 26 (6.244997998) | 27.5 (12.02081528) | 26.6 (7.503332593)
The Delis Kaplan Color Word Interference Test, inhibition [Mean (Standard Deviation); unit: Time - seconds] — Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 150 (maximum). Longer time indicates worse performance. is 0-150 seconds. Longer time indicates worse performance.
  Time - seconds | 57 (5) | 71.5 (9.192388155) | 62.8 (9.833615815)
The Delis Kaplan Color Word Interference Test, inhibition and switching [Mean (Standard Deviation); unit: Time - seconds] — Evaluation of the Delis Kaplan Color Word Interference Test. Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 240 (maximum). Longer time indicates worse performance.
  Time - seconds | 71.33333333 (19.85782801) | 75 (16.97056275) | 72.8 (16.52876281)
Rey Auditory Verbal Learning Test and alternative lists, total learning [Mean (Standard Deviation); unit: Total items] — Evaluation of Rey Auditory Verbal Learning Test. Metric: Number of Total learning items and Correct Recalls. Total Range 0 (minimum) - 75 (maximum). Larger numbers indicate better performance.
  Total items | 40.66666667 (15.14375559) | 48.5 (3.535533906) | 43.8 (11.67047557)
Rey Auditory Verbal Learning Test and alternative lists, delayed recall [Mean (Standard Deviation); unit: Total items] — Evaluation of treatment differences (active versus sham) in change in Rey Auditory Verbal Learning Test. Metric: Total Number of Delayed Recall items and Correct Recalls. Total Range 0 (minimum) - 15 (maximum). Larger numbers indicate better performance.
  Total items | 7.333333333 (5.033222957) | 9.5 (0.707106781) | 8.2 (3.768288736)

OUTCOME MEASURES:

1. Primary Outcome: The Controlled Oral Word Association Test
Description: Evaluation of treatment differences (active versus sham) in change on the Control Word Association Test. Metric: Total Number of Correct Items Generated for three different letters. Total Range 0 (minimum) - 200 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: n=3 assigned to Active to Sham arm completed phase 1 (Baseline, Immediately post phase 1 intervention, 8 weeks after post phase 1 intervention), and only n=2 assigned to Active to Sham arm completed phase 2 (Immediately post phase 2 intervention, 8 weeks after post phase 2 intervention). n=2 assigned to Sham to Active completed both phases 1 &2.
Measure: Mean (Standard Deviation); unit: Total items
Groups:
- Active to Sham: Subjects in this arm were first randomly assigned to receive active stimulation. After completion of active stimulation, subjects were assigned to sham stimulation.
- Sham to Active: Subjects in this arm were first randomly assigned to receive sham stimulation. After completion of active stimulation, subjects were assigned to active stimulation.
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 30.67 (7.23) | 30.5 (0.71)
  Immediate post completion of phase 1 intervention | 33.33 (5.69) | 35 (0)
  8 weeks post completion of phase 1 intervention | 34.67 (7.51) | 39.5 (7.78)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  Immediate post completion of phase 2 intervention | 31 (9.9) | 48.5 (3.54)
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 33.5 (4.95) | 43.5 (4.95)

2. Primary Outcome: Category Fluency
Description: Evaluation of treatment differences (active versus sham) in change on Category Fluency. Metric: Total Number of Correct Items Generated for Animal. Total Range 0 (minimum) - 100 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 18 (1.73) | 17 (0)
  Immediate post completion of phase 1 intervention | 17.67 (6.35) | 24.5 (0.71)
  8 weeks post completion of phase 1 intervention | 20 (2.65) | 22.5 (0.71)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  Immediate post completion of phase 2 intervention | 11 (1.41) | 27.5 (3.54)
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 17.5 (2.12) | 20.5 (0.71)

3. Primary Outcome: The Boston Naming Test
Description: Evaluation of treatment differences (active versus sham) in change on The Boston Naming Test - 30 items. Metric: Total Number of Correct Items Generated. Total Range 0 (minimum) - 30 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: n=3 assigned to Active to Sham arm completed phase 1 (Baseline, Immediately post phase 1 intervention, 8 weeks after post phase 1 intervention), and only n=2 assigned to Active to Sham arm completed phase 2 (Immediately post phase 2 intervention, 8 weeks after post phase 2 intervention).
  n=2 assigned to Sham to Active completed both phases 1 &2, except for one subject in the Sham to Active group missed data at the immediate post time point for phase 2.
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 26.67 (2.52) | 28 (0)
  Immediate post completion of phase 1 intervention | 27 (1) | 29.5 (0.71)
  8 weeks post completion of phase 1 intervention | 27.33 (1.53) | 28.5 (2.12)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 27 (1.41) | 30 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 28 (2.83) | 30 (0)

4. Primary Outcome: Semantic Object Retrieval Test
Description: Evaluation of treatment differences (active versus sham) in change in Semantic Object Retrieval Test. Metric: Total Number of Correct Retrievals. Total Range 0 (minimum) - 32 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 30.33 (1.53) | 30.5 (2.12)
  Immediate post completion of phase 1 intervention | 31.33 (1.15) | 31.5 (0.71)
  8 weeks post completion of phase 1 intervention | 30.67 (1.15) | 31 (1.41)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 30 (1.41) | 31 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 32 (0) | 31.5 (0.71)

5. Primary Outcome: The Delis Kaplan Color Word Interference Test, Naming
Description: Evaluation of treatment differences (active versus sham) in change on the Delis Kaplan Color Word Interference Test. Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 150 (maximum). Longer time indicates worse performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 35.66666667 (5.131601439) | 41 (7.071067812)
  Immediate post completion of phase 1 intervention | 32.66666667 (2.516611478) | 31 (8.485281374)
  8 weeks post completion of phase 1 intervention | 31.66666667 (4.509249753) | 34.5 (7.778174593)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 34.5 (3.535533906) | 32 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 29 (5.656854249) | 34.5 (3.535533906)

6. Primary Outcome: The Delis Kaplan Color Word Interference Test, Reading
Description: as for outcome 5
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 26 (6.244997998) | 27.5 (12.02081528)
  Immediate post completion of phase 1 intervention | 24 (7) | 24 (4.242640687)
  8 weeks post completion of phase 1 intervention | 25.66666667 (6.658328118) | 25.5 (7.778174593)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 31.5 (3.535533906) | 27 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 24.5 (0.707106781) | 27 (4.242640687)

7. Secondary Outcome: The Trail Making Test - Part A
Description: Evaluation of treatment differences (active versus sham) in change on the Trail Making Test (Parts A&B). Metric: Time to Solution. Total Range 0 (minimum) - 300 (maximum). Longer time indicates worse performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 37.66666667 (14.36430762) | 41.5 (7.778174593)
  Immediate post completion of phase 1 intervention | 27.66666667 (11.93035345) | 26.5 (13.43502884)
  8 weeks post completion of phase 1 intervention | 28 (19.28730152) | 27 (5.656854249)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 30.5 (14.8492424) | 29 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 34.5 (26.1629509) | 26.5 (9.192388155)

8. Secondary Outcome: The Trail Making Test - Part B
Description: as for outcome 7
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 68.66666667 (21.57158625) | 101 (9.899494937)
  Immediate post completion of phase 1 intervention | 63.66666667 (3.511884584) | 52.5 (16.26345597)
  8 weeks post completion of phase 1 intervention | 57.66666667 (21.22105872) | 63.5 (7.778174593)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 61.5 (10.60660172) | 62 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 58 (15.55634919) | 71.5 (7.778174593)

9. Secondary Outcome: Digit Span Forward
Description: Evaluation of treatment differences (active versus sham) in change in Digit Span Forward. Metric: Memory Span, a composite score of how many numbers are repeated correctly in a forward order. Z = 0 is the normed average, with positive Z values better and negative Z values worse than the normed average.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Z scale
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Units on Z scale
  Baseline | 0.933333333 (1.078579312) | 0.4 (0.707106781)
  Immediate post completion of phase 1 intervention | 0.3 (0.556776436) | -0.085 (0.021213203)
  8 weeks post completion of phase 1 intervention | -0.34 (0.819023809) | -0.1 (0)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 0.05 (0.494974747) | -1.05 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | -0.85 (0.777817459) | -0.575 (0.671751442)

10. Secondary Outcome: Digit Span Backward
Description: Evaluation of treatment differences (active versus sham) in change in Digit Span Backward. Metric: Memory Span, a composite score of how many numbers are repeated correctly in a backward order. Z = 0 is the normed average, with positive Z values better and negative Z values worse than the normed average.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Z scale
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Units on Z scale
  Baseline | 0.2 (1.252996409) | 0.7 (1.272792206)
  Immediate post completion of phase 1 intervention | -0.933333333 (0.56862407) | 1.525 (0.035355339)
  8 weeks post completion of phase 1 intervention | 0.44 (0.991362699) | 0.25 (0.636396103)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 0.81 (1.965756852) | -0.19 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 0.385 (2.566797616) | 0.68 (0.028284271)

11. Primary Outcome: The Delis Kaplan Color Word Interference Test, Inhibition
Description: as for outcome 5
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 57 (5) | 71.5 (9.192388155)
  Immediate post completion of phase 1 intervention | 46 (2.645751311) | 64 (9.899494937)
  8 weeks post completion of phase 1 intervention | 53 (3.464101615) | 58.5 (9.192388155)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 48 (5.656854249) | 66 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 46.5 (0.707106781) | 59.5 (2.121320344)

12. Primary Outcome: The Delis Kaplan Color Word Interference Test, Inhibition and Switching
Description: Evaluation of treatment differences (active versus sham) in change on the Delis Kaplan Color Word Interference Test. Metric: Time - seconds to Name Items. Total Range 0 (minimum) - 240 (maximum). Longer time indicates worse performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Time - seconds
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Time - seconds
  Baseline | 71.33333333 (19.85782801) | 75 (16.97056275)
  Immediate post completion of phase 1 intervention | 72 (29.13760457) | 58 (8.485281374)
  8 weeks post completion of phase 1 intervention | 75.33333333 (24.19366308) | 56.5 (6.363961031)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 61.5 (3.535533906) | 53 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 70 (9.899494937) | 52 (0)

13. Primary Outcome: Rey Auditory Verbal Learning Test and Alternative Lists, Total Learning
Description: Evaluation of treatment differences (active versus sham) in change in Rey Auditory Verbal Learning Test. Metric: Number of Total learning items and Correct Recalls. Total Range 0 (minimum) - 75 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 40.66666667 (15.14375559) | 48.5 (3.535533906)
  Immediate post completion of phase 1 intervention | 39.33333333 (11.8462371) | 57 (7.071067812)
  8 weeks post completion of phase 1 intervention | 43.66666667 (11.59022577) | 58 (4.242640687)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 40.5 (17.67766953) | 73 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 38.5 (3.535533906) | 63 (7.071067812)

14. Primary Outcome: Rey Auditory Verbal Learning Test and Alternative Lists, Delayed Recall
Description: Evaluation of treatment differences (active versus sham) in change in Rey Auditory Verbal Learning Test. Metric: Total Number of Delayed Recall items and Correct Recalls. Total Range 0 (minimum) - 15 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 7.333333333 (5.033222957) | 9.5 (0.707106781)
  Immediate post completion of phase 1 intervention | 6 (4.582575695) | 12 (1.414213562)
  8 weeks post completion of phase 1 intervention | 8.666666667 (4.509249753) | 13.5 (2.121320344)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 7.5 (6.363961031) | 15 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 7 (1.414213562) | 11.5 (3.535533906)

15. Secondary Outcome: Rey-Osterrieth Complex Figure Test - Delayed Recall
Description: Evaluation of treatment differences (active versus sham) in change in Rey-Osterrieth Complex Figure Test scores. Metric: Score. Total Range 0 (minimum) - 36 (maximum). This is a summed score of the number and accuracy of complex figure features captured. Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 15.16666667 (0.577350269) | 25.5 (2.121320344)
  Immediate post completion of phase 1 intervention | 18.5 (3.905124838) | 28 (9.899494937)
  8 weeks post completion of phase 1 intervention | 18 (5.408326913) | 32.5 (0.707106781)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 14 (9.899494937) | 31 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 24 (11.3137085) | 25.45 (3.606244584)

16. Secondary Outcome: The Digit Symbol Substitution Test
Description: Evaluation of treatment differences (active versus sham) in change on the Digit Symbol Substitution Test. Metric: Number of Items. Total Range 0 (minimum) - 135 (maximum). Larger numbers indicate better performance.
Time Frame: Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Total items
Arm/Group | Active to Sham | Sham to Active
Number analyzed (Participants) | 3 | 2
Total items
  Baseline | 45 (5.196152423) | 45.5 (14.8492424)
  Immediate post completion of phase 1 intervention | 45.33333333 (2.516611478) | 58 (11.3137085)
  8 weeks post completion of phase 1 intervention | 47.66666667 (1.527525232) | 58.5 (23.33452378)
  Immediate post completion of phase 2 intervention: number analyzed (Participants) | 2 | 1
  Immediate post completion of phase 2 intervention | 50 (4.242640687) | 53 (NA) — Only one subject
  8 weeks post completion of phase 2 intervention: number analyzed (Participants) | 2 | 2
  8 weeks post completion of phase 2 intervention | 48 (4.242640687) | 62.5 (9.192388155)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 8 weeks
Arm/Group | Active to Sham Transcranial Direct Current Stimulation | Sham to Active Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT05408975/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT05408975/ICF_001.pdf